CLINICAL TRIAL: NCT01094821
Title: A Double Blind, Randomized, Placebo Controlled, Parallel Group Study to Investigate the Effect of ATI-7505 on Gastric Emptying and Small Bowel and Colonic Transit in Healthy Volunteers
Brief Title: Effect of ATI-7505 on Gastrointestinal Transit in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: ARYx Therapeutics (Industry)
Responsible Party: Michael Camilleri, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB 276-05; IND 68,208 (Other: FDA issued IND number)
Record Dates: First submitted 2009-08-04; First posted 2010-03-29 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Healthy
Keywords: Healthy volunteers; ATI-7505; Scintigraphy; Gastrointestinal transit
MeSH Terms: interventions — ATI 7505

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 3 mg ATI-7505 (Experimental): 3 mg ATI-7505 three times daily for 9 days followed by transit scintigraphy
  Interventions: Drug: ATI-7505
- Placebo (Placebo Comparator): Placebo capsule three times daily for 9 days followed by transit scintigraphy
  Interventions: Drug: Placebo
- 10 mg ATI-7505 (Experimental): 10 mg ATI-7505 three times daily for 9 days followed by transit scintigraphy
  Interventions: Drug: ATI-7505
- 20 mg ATI-7505 (Experimental): 20 mg ATI-7505 three times daily for 9 days followed by transit scintigraphy
  Interventions: Drug: ATI-7505

INTERVENTIONS:
Drug: ATI-7505 — 3 mg three times daily for 9 days
  Arms: 3 mg ATI-7505
Drug: Placebo — Placebo capsule three times daily for 9 days
  Arms: Placebo
Drug: ATI-7505 — 10 mg ATI-7505 three times daily for 9 days
  Arms: 10 mg ATI-7505
Drug: ATI-7505 — 20 mg ATI-7505 three times daily for 9 days
  Arms: 20 mg ATI-7505

SUMMARY:
This is a pharmacodynamic study in healthy volunteers to determine the effects of a new 5-HT4 agonist on gastric, small bowel and colonic transit.

DETAILED DESCRIPTION:
ATI-7505, is an engineered analog of the 5-HT4 agent, cisapride. The objectives of this study are to compare effects of ATI-7505 and placebo on gastric, small bowel and colonic transit in healthy human volunteers and evaluate the safety and tolerability of ATI-7505.

This trial is a double-blind, randomized, placebo-controlled study evaluating the gastrointestinal transit effects of ATI-7505 and placebo. Three different doses (3, 10, 30mg) of ATI-7505 and placebo will be administered in parallel to four independent groups of 12 subjects each. The maximum duration of drug exposure for any subject is 9 days.

All participants will undergo a standard 48 hour gastrointestinal transit measurement using scintigraphy with standardized meals during the first 12 hours. The response endpoints (colonic geometric center at 4 h, colonic geometric center at 24 h, colonic geometric center at 48 h, gastric residual at 2 & 4 h, colonic filling at 6 h and ascending colonic emptying t1/2) will be based on abdominal scintigraphic images following the technetium-99m egg meal and methacrylate-coated, delayed-release capsule containing 111In labeled activated charcoal.

Safety and tolerability will be evaluated by serial assessment of vital signs, physical examination, ECG, adverse events, concomitant medications and blood sample analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers between the ages of 18 to 65 years old (inclusive) with a BMI ≥ 18 and ≤ 32
2. PR, QRS and QT intervals within normal limits on screening ECG. Specifically, PR < 220 msec, QRS < 140 msec, QTc < 450 msec
3. Are able and willing to understand study requirements, follow instructions, attend all required study visits (especially during 48 hrs of scintigraphic scan), undergo all planned tests (including drawing of blood samples and consumption of standardized study meals)
4. Are able and willing to sign IRB-approved, written informed consent to participate in this study
5. Have had negative urine screen and clinical history (prior 2 years) for drugs of abuse at screening visit
6. Women with no child bearing potential, as defined by at least 1 year post-menopausal (absence of vaginal bleeding or spotting) or surgically sterile. Men will have a sterile sexual partner or will, starting at time of study drug administration a minimum of 1 month after study drug administration, be willing to use an approved method of contraception (which may include use of a condom with spermicide or use by partner of oral, implantable or injectable contraceptives, IUD, diaphragm with spermicide)

Exclusion Criteria

1. Inability to understand study requirements or follow study procedures (especially entire 48 h of scintigraphy examination), attend all required study visits, undergo all planned tests (including drawing of blood samples and consumption of study meals)
2. Any out of range laboratory value at screening that has not been reviewed, approved and documented as not clinically significant (NCS) by the Principal Investigator.
3. Use of alcohol within 24 h of randomization visit (Visit 2) and through completion of the study
4. History of untoward effects of metoclopramide
5. Any clinically significant abnormality on screening ECG.
6. Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Principal Investigator, would make the subject unsuitable for the study or put them at additional risk)
7. Known allergy, hypersensitivity or sensitivity to cisapride
8. Pregnancy or lactation
9. History of alcohol or other substance abuse within the past two years
10. Received treatment with any other investigational drug within the preceding 30 days or 5 half-lives, whichever is greater
11. Major surgery within 3 months of study entry and any surgery within 2 weeks of study entry unless approved by the Principal Investigator and Sponsor?s Medical Monitor
12. Any documented history of irregular intestinal transit including but not limited to gastro-esophageal reflux disease (GERD), gastroparesis of any kind, irritable bowel syndrome, inflammatory bowel disease and chronic constipation or diarrhea under the care of a physician and/or requiring daily medication
13. Any history of gastrointestinal tract or abdominal surgery, except tubal ligation, hysterectomy, appendectomy, cholecystectomy or hemorrhoid surgery > 3 months prior to screening
14. More than three positive (i.e., ?yes?) responses on screening bowel symptom questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Colonic geometric center at 24 h | 24 hours
  Colonic geometric center determined 24 hours post first camera image following ingestion of study medication with Indium-111 capsule and breakfast with Technetium-99 labeled egg breakfast
Ascending colonic emptying t1/2 | 24 hours
  As measured with scintigraphic method following 111In labeled capsule and 99Tc labeled egg breakfast
Gastric emptying of solids (T1/2) | 4 hours
  As measured with scintigraphic method following technetium-99m egg meal

SECONDARY OUTCOMES:
Colonic filling at 6 h | 6 hours
  As measured with scintigraphic method following ingestion of 111In labeled capsule and 99Tc labeled egg breakfast
Colonic geometric center at 48 hours | 48 hours
  As measured with scintigraphic method following ingestion of In111 capsule and Tc99 labeled breakfast
Percent gastric emptying at 1, 2 and 4 hours | 4 hours
  As measured with scintigraphic method following ingestion of 99Tc labeled egg breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Camilleri M, Vazquez-Roque MI, Burton D, Ford T, McKinzie S, Zinsmeister AR, Druzgala P. Pharmacodynamic effects of a novel prokinetic 5-HT receptor agonist, ATI-7505, in humans. Neurogastroenterol Motil. 2007 Jan;19(1):30-8. doi: 10.1111/j.1365-2982.2006.00865.x. PMID 17187586